CLINICAL TRIAL: NCT04873440
Title: A Phase I/II, Open-label Study to Evaluate the Abscopal Response and Safety of Manganese and Standard-of-care Radiotherapy/ SBRT in Subjects With Metastatic Solid Tumors or Lymphoma
Brief Title: An Open-label, Phase I/II Study of Manganese Plus Radiotherapy in Patients With Metastatic Solid Tumors or Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-063
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumor; Lymphoma
Keywords: metastatic; radiotherapy; manganese; abscopal response
MeSH Terms: conditions — Lymphoma; Neoplasm Metastasis | interventions — manganese chloride; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manganese plus Radiotherapy (Experimental): Subject received standard-of-care radiotherapy or stereotactic body radiation therapy (SBRT) to one metastatic site. Manganese inhalation began 1 week after the start of radiotherapy and lasted up to 6 months. The same systemic therapy before the enrollment will be maintained.
  Interventions: Drug: Manganese Chloride; Radiation: Radiotherapy; Drug: Chemo-immunotherapy

INTERVENTIONS:
Drug: Manganese Chloride — Administered by inhalation at 0.4mg/kg/d twice a week
  Other Names: Mn2+
Radiation: Radiotherapy — Measurable lesions were targeted for radiotherapy at the discretion of the treating physician.Standard-of-care radiotherapy or SBRT were both allowed.
Drug: Chemo-immunotherapy — The same chemotherapy and/or anti-PD-1 therapy before thei patients' enrolment were allowed. Whether and which should be given depends on the treatment regimen before enrollment.

SUMMARY:
Radiotherapy is a regular care for metastatic solid tumors or lymphoma, and it can induce immunogenic death of tumor cells and a stronger immune response. Sometimes, tumor regression would be observed at sites distant to an irradiated field because of the radiotherapy-induced anticancer immune responses, so-called abscopal response. Manganese has been confirmed to activate innate immune and function as anticancer immunoadjuvant in pre-clinical studies. This study is designed to assess the abscopal response and safety of combined therapy of manganese and radiotherapy in patients with metastatic solid tumors or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically proven metastatic solid tumors or lymphoma.
2. Subjects must have at least two distinct measurable sites of disease (≥1 cm).
3. ≥ 18 years old.
4. Life expectancy of at least 6 months.
5. Eastern Cooperative Oncology Group performance status 0-2.
6. Subjects must have stable or progressing disease to the ongoing systemic therapy.
7. Multiple lines of previous chemo-immunotherapy were permitted.
8. Patients with known brain metastases were included in the trial but brain lesions were not eligible as target or non-target lesions.
9. Adequate organ function.
10. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.
11. Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Prior organ allograft.
4. Women who are pregnant or breastfeeding.
5. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
6. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
7. Subjects with previous or concurrent other malignancies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-06 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with an abscopal response | 6 months
  An abscopal response was defi ned as a decrease in the longest diameter of at least 30% in any measurable (≥1 cm) non-irradiated lesion from baseline.
Number of subjects with treatment-related adverse events (AEs) | 12 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. AEs were considered to be treatment-related if they had started or worsened within the interval from first study drug administration until the follow-up visit.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 12 months
  DCR is defined as the proportion of subjects who achieved a stable disease (SD), partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression-free survival (PFS) | 24 months
  PFS time was measured from study entry to the first documentation of disease progression or death. Disease progression was determined per the RECIST V1.1.
Overall survival (OS) | 24 months
  OS time was measured from the study entry to the date of death.
Number of participants with laboratory test abnormalities | 12 months
  The laboratory tests of serum cytokines and chemokines will be performed on day 1 and 3 of each cycle, and the abnormality will be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided